CLINICAL TRIAL: NCT02256345
Title: Pharmacokinetics, Pharmacodynamics, and Impact of Inorganic Nitrate on Exercise in HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01340
Record Dates: First submitted 2014-09-30; First posted 2014-10-03 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-08

CONDITIONS: Heart Failure; Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic | interventions — potassium nitrate; Potassium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- KNO3 active comparator (Active Comparator): KNO3 will be given at a dose of 6 mmol twice daily for the first week, increasing to 6 mmol three times daily for the second week if well tolerated
  Interventions: Drug: KNO3
- KCl placebo comparator (Placebo Comparator): KCl will be used as a placebo and will be given as 6 mmol twice daily for the first week, increasing to 6 mmol three times daily for the second week if well tolerated
  Interventions: Drug: KCl

INTERVENTIONS:
Drug: KNO3 — Active Comparator
  Other Names: Potassium Nitrate
  Arms: KNO3 active comparator
Drug: KCl — Placebo Comparator
  Other Names: Potassium Chloride
  Arms: KCl placebo comparator

SUMMARY:
This study will be performed to determine the safety, tolerability, and dose-response to inorganic nitrate on exercise capacity in HFpEF. There are two primary goals for this study:

1. Determine the population-specific pharmacokinetics and dose of KNO3 that can be safely given to subjects with HFpEF.
2. Determine if there is a dose-response effect of nitrate supplementation on exercise capacity, evidenced by peak oxygen consumption (peak VO2), and physiologic adaptations to exercise.

DETAILED DESCRIPTION:
This study randomized subjects to either placebo (n=3) or KNO3 (n=9) given a sequential dosing regimen: 6 mmol twice daily for 1 week followed by dose escalation to 6 mmol thrice daily for 1 week). Although a primary goal of the study was to assess the safety of KNO3 and within-group changes in various end points in KNO3-treated subjects, a small number of placebo-treated (PB, n=3) subjects were included only to assess for any potential training effect on repeated exercise and Kansas City Cardiomyopathy Questionnaire (KCCQ) measurements. Potassium chloride, given in equivalent doses, was used as the PB to account for differences in blood pressure or flow that could be attributed to potassium.

The study was initially designed to be single-blinded to allow the principal investigator to be aware of arm allocation because of potential concerns for methemoglobinemia with drug administration. One investigator, who was the primary investigator responsible for supervising all visits and measurements during the study, remained blinded to treatment allocation throughout the entirety of the study. All physiological and imaging data were analyzed in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA Class II-III symptoms.
2. LV EF > 50%.
3. Stable medical therapy for at least 1 month.
4. Evidence of significant diastolic dysfunction, meeting the European Society of Echocardiography criteria for HFpEF.

Exclusion Criteria

1. Any rhythm other than sinus with native conduction.
2. Inability to exercise.
3. Moderate or greater valvular disease.
4. Hypertrophic, infiltrative, or inflammatory cardiomyopathy.
5. Pericardial disease.
6. Current angina.
7. Acute coronary syndrome or coronary intervention within the past 2 months.
8. Primary pulmonary arteriopathy.
9. Clinically significant lung disease.
10. Ischemia on stress testing without subsequent revascularization.
11. Treatment with phosphodiesterase inhibitors that cannot be withheld.
12. Treatment with organic nitrates or allopurinol.
13. Significant liver disease impacting synthetic function or volume control.
14. Poor echocardiographic windows.
15. eGFR < 30 mL/min/m2 or Cr >2.5.
16. Current smoking.
17. Alcohol dependency.
18. History of Barret's esophagus.
19. G6PD deficiency
20. Methemoglobinemia - baseline methemoglobin level >3% prior to any study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio A Chirinos, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Zamani P, Tan V, Soto-Calderon H, Beraun M, Brandimarto JA, Trieu L, Varakantam S, Doulias PT, Townsend RR, Chittams J, Margulies KB, Cappola TP, Poole DC, Ischiropoulos H, Chirinos JA. Pharmacokinetics and Pharmacodynamics of Inorganic Nitrate in Heart Failure With Preserved Ejection Fraction. Circ Res. 2017 Mar 31;120(7):1151-1161. doi: 10.1161/CIRCRESAHA.116.309832. Epub 2016 Dec 7. PMID 27927683

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized to KNO3: KNO3 will be given at a dose of 6 mmol twice daily for the first week, increasing to 6 mmol three times daily for the second week if well tolerated.
  Active Comparator: Potassium Nitrate (KNO3)
- Randomized to KCl: KCl will be used as a placebo and will be given as 6 mmol twice daily for the first week, increasing to 6 mmol three times daily for the second week if well tolerated.
  Placebo Comparator: Potassium Chloride (KCl)
Period: Overall Study
Arm/Group | Randomized to KNO3 | Randomized to KCl
Started | 9 | 3
Completed | 9 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized to KNO3: KNO3 will be given at a dose of 6 mmol twice daily for the first week, increasing to 6 mmol three times daily for the second week if well tolerated
  Active Comparator: Potassium Nitrate
- Randomized to KCl: KCl will be used as a placebo and will be given as 6 mmol twice daily for the first week, increasing to 6 mmol three times daily for the second week if tolerating well.
  Placebo Comparator: Potassium Chloride
- Total: Total of all reporting groups
Arm/Group | Randomized to KNO3 | Randomized to KCl | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (5.5) | 62.7 (8.0) | 62.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, n (%): White | 5 | 3 | 8
  Race, n (%): Black | 3 | 0 | 3
  Race, n (%): Pacific Islander | 1 | 0 | 1
New York Heart Association Heart failure classification (NYHA Class) n (%) [Count of Participants; unit: Participants] — Class II- Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea (shortness of breath).
  Class III- Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Participants
    Class II | 8 | 2 | 10
    Class III | 1 | 1 | 2
Body Mass Index, kg/m^2, mean (SD) [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (6.3) | 37.4 (9.9) | 34.4 (7.0)
Number of Obese Participants, n(%) [Count of Participants; unit: Participants] | 5 | 3 | 8
Number of Hypertensive Participants, n(%) [Count of Participants; unit: Participants] | 9 | 3 | 12
Number of Participants with Hyperlipidemia, n (%) [Count of Participants; unit: Participants] | 7 | 3 | 10
Number of Participants with Coronary Artery Disease, n (%) [Count of Participants; unit: Participants] | 3 | 1 | 4
Number of Participants with History of atrial fibrillation, n (%) [Count of Participants; unit: Participants] | 0 | 1 | 1
Number of Participants with Diabetes Mellitus, n (%) [Count of Participants; unit: Participants] | 5 | 2 | 7
Number of Participants with Obstructive sleep apnea, n (%) [Count of Participants; unit: Participants] | 3 | 3 | 6
Number of Participants with Current Continuous Positive Airway Pressure (CPAP) use, n (%) [Count of Participants; unit: Participants] | 2 | 3 | 5
Number of Participants with Obstructive lung disease, n (%) [Count of Participants; unit: Participants] | 2 | 1 | 3
Number of Participants on Beta-blockers, n (%) [Count of Participants; unit: Participants] | 7 | 2 | 9
Number of Participants onACEI/ARB, n (%) [Count of Participants; unit: Participants] | 7 | 2 | 9
Number of Participants on Mineralocorticoid receptor antagonists, n (%) [Count of Participants; unit: Participants] | 2 | 1 | 3
Number of Participants on Calcium-channel blockers, n (%) [Count of Participants; unit: Participants] | 3 | 1 | 4
Number of Participants on Loop diuretics, n (%) [Count of Participants; unit: Participants] | 7 | 2 | 9
Number of Participants on Thiazide diuretic, n (%) [Count of Participants; unit: Participants] | 3 | 1 | 4
Number of Participants on Statin, n (%) [Count of Participants; unit: Participants] | 5 | 2 | 7
Estimated Glomerular Filtration Rate (eGFR), mL/min per 1.73m^2, mean (SD) [Mean (Standard Deviation); unit: mL/min per 1.73m^2] | 71.0 (14.1) | 64.7 (5.9) | 69.4 (12.6)
Estimated Glomerular Filtration Rate (eGFR) <60 mL/min per 1.73m^2, n (%) [Count of Participants; unit: Participants] | 3 | 1 | 4
N-terminal pro-brain natriuretic peptide (NT-proBNP), pg/ml, mean (SD) [Mean (Standard Deviation); unit: pg/ml] | 108.3 (94.7) | 119 (87.0) | 111 (89.0)
Number of Participants with high N-terminal pro-brain natriuretic peptide (NT-proBNP), pg/ml, n (%) [Count of Participants; unit: Participants] | 3 | 2 | 5
Hemoglobin, g/dL, mean (SD) [Mean (Standard Deviation); unit: g/dL] | 13.6 (0.8) | 13.5 (1.0) | 13.6 (0.8)
Methemoglobin, %, mean (SD) [Mean (Standard Deviation); unit: percent of total hemoglobin] | 1.0 (0.2) | 1.0 (0.5) | 1.0 (0.3)
Left Ventricular (LV) mass,g, mean (SD) [Mean (Standard Deviation); unit: g] | 174.43 (77.09) | 165.98 (19.27) | 172.32 (66.36)
Left Ventricular (LV) mass index, g/m^2, mean (SD) [Mean (Standard Deviation); unit: g/m^2] | 79.78 (26.01) | 76.18 (7.33) | 78.88 (22.46)
Relative wall thickness, mean (SD) [Mean (Standard Deviation); unit: ratio] — The ratio of twice LV diastolic posterior wall thickness to left ventricular end-diastolic dimension
  ratio | 0.47 (0.09) | 0.46 (0.09) | 0.47 (0.09)
Mitral early inflow velocity (E), cm/s, mean (SD) [Mean (Standard Deviation); unit: cm/s] | 74.53 (24.75) | 85.73 (7.04) | 77.33 (21.91)
Mitral atrial inflow velocity (E), cm/s, mean (SD) [Mean (Standard Deviation); unit: cm/s] | 70.74 (20.06) | 88.61 (21.28) | 75.21 (20.99)
Septal tissue doppler early velocity (e'), mm/s, mean (SD) [Mean (Standard Deviation); unit: mm/s] | 70.64 (12.45) | 93.71 (28.65) | 76.41 (19.26)
Septal E/e' ratio, mean (SD) [Mean (Standard Deviation); unit: ratio] | 10.70 (3.76) | 9.60 (2.39) | 10.42 (3.40)
Left atrial volume index, mL/m^2, mean (SD) [Mean (Standard Deviation); unit: mL/m^2] | 27.20 (7.87) | 29.38 (5.33) | 27.74 (7.15)
Left ventricular ejection fraction, %, mean (SD) [Mean (Standard Deviation); unit: % (stroke volume/ end-diastolic vol)x100] | 65.84 (7.74) | 59.41 (13.66) | 64.23 (9.27)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Uptake (VO2) From Baseline Upto 1 Week of Administration for Each Dose
Description: Peak oxygen uptake (VO2) defined as the average value obtained during the last 30 seconds of exercise.
Time Frame: Baseline, end of week 1, end of week 2
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Randomized to KNO3 | Randomized to KCl
Number analyzed (Participants) | 9 | 3
L/min
  Baseline Viist | 1.16 [1.13 to 1.19] | 1.49 [1.43 to 1.54]
  End of week 1 visit | 1.20 [1.17 to 1.24] | 1.44 [1.39 to 1.49]
  End of week 2 visit | 1.20 [1.17 to 1.23] | 1.44 [1.39 to 1.50]

2. Secondary Outcome: Change in Vasodilatory Reserve for Each Dose
Description: Percent change in peak vascular resistance from rest to peak exercise
Time Frame: Baseline, end of week 1, end of week 2
Measure: Mean (95% Confidence Interval); unit: %change in peak vascular resistance
Arm/Group | Randomized to KNO3 | Randomized to KCl
Number analyzed (Participants) | 9 | 3
%change in peak vascular resistance
  Baseline | -25.6 [-40.9 to -10.4] | -25.8 [-31.4 to -20.3]
  End of week 1 visit | -27.1 [-43.6 to -10.5] | -30.6 [-36.2 to -25.1]
  End of week 2 visit | -34.2 [-49.4 to -18.9] | -20.0 [-24.2 to -15.8]

3. Secondary Outcome: Change in Mitochondrial Oxidative Capacity for Each Dose
Description: Percent change in oxidative capacity (oxyhemoglobin levels) before and after occlusion
Time Frame: Baseline, end of week 1, end of week 2
Measure: Mean (95% Confidence Interval); unit: Percent change in oxidative capacity
Arm/Group | Randomized to KNO3 | Randomized to KCl
Number analyzed (Participants) | 9 | 3
Percent change in oxidative capacity
  Baseline | 63.2 [47.6 to 78.8] | 106.5 [59.2 to 153.7]
  End of week 1 visit | 59.2 [42.1 to 76.2] | 110.4 [63.2 to 157.7]
  End of Week 2 visit | 62.2 [46.6 to 77.7] | 45.4 [5.0 to 85.8]

4. Secondary Outcome: Change in Aortic Augmentation Index
Description: Percent change in augmentation index, whereas augmentation index at each time point (visit) is defined as the amplitude of the second peak to the first peak of the aortic pulse wave form multiplied by 100: augmentation index = (P2/P1)×100.
Time Frame: Baseline, end of week 1, end of week 2
Measure: Mean (95% Confidence Interval); unit: Percent change in augumentation index
Arm/Group | Randomized to KNO3 | Randomized to KCl
Number analyzed (Participants) | 9 | 3
Percent change in augumentation index
  Baseline visit | 3.0 [-5.4 to 11.4] | -2.3 [-11.5 to 6.8]
  End of week 1 visit | -5.4 [-13.1 to 2.4] | -11.9 [-23.5 to -0.2]
  End of week 2 visit | -7.1 [-14.9 to 0.6] | -0.2 [-9.4 to 9.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at every visit. There are a total of three visits that are 1 week apart.
Description: All adverse events were non serious so they are reported under Other Adverse Events
Arm/Group | Randomized to KNO3 | Randomized to KCl
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 5/9 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to KNO3 (N=9) | Randomized to KCl (N=3)
Any side effect (General disorders) | 4 | 1 (1)
GI symptoms (Gastrointestinal disorders) | 3 | 1 — Includes GI upset, nausea, vomiting, flatulence
Headache (Nervous system disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Mild lower extremity edema (Cardiac disorders) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
* Small sample size
* Serial blood draws, which caused a decrease in hemoglobin concentration, which may have constrained the increase in VO2,peak and reduced the magnitude of the improvement in exercise capacity and quality of life.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No